CLINICAL TRIAL: NCT03073538
Title: Screening of Gonococcal and Chlamydial Infections in the Third Trimester
Status: Completed | Type: Observational
Sponsor: Unity Health Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: 16-337
Record Dates: First submitted 2017-02-15; First posted 2017-03-08 (Actual); Last update posted 2019-02-21 (Actual); Status verified 2019-02

CONDITIONS: Gonococcal Infection; Chlamydia Infections
MeSH Terms: conditions — Gonorrhea; Chlamydia Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Untreated maternal infection with gonorrhea and/or chlamydia can have serious complications in pregnancy and the neonatal period. In Ontario, routine screening for these infections is done in the first trimester of pregnancy, positive cases are treated with antibiotics, and all newborns are given antibiotic eye ointment within 24 hours of birth. Recently, the Canadian Pediatric Society recommended stopping universal prophylaxis for newborns, with instead, focus on screening and treatment of these infections in pregnancy. Given that these infections can occur at any time in pregnancy, and exposure at delivery provides a significant risk to infants, more information is needed about the rates of infection throughout pregnancy and health-care provider compliance with guidelines to make this change without undue risk. With this information optimal timing of testing can be evaluated.

DETAILED DESCRIPTION:
The primary objective of this study is to retrospectively examine the incidence rates of N. gonorrhoeae (NG) and C. trachomatis (CT) in the first and third trimester for the obstetrical population at St. Michael's Hospital over the course of six months. Secondary objectives include (1) feasibility of instituting third trimester screening for sexually transmitted infections, and (2) assessment of physician compliance with Canadian screening and treatment guidelines. This information will help us to deduce the optimal timing of screening for NG and CT in the obstetrical population at St. Michael's Hospital.

It is hypothesized that the incidence rates of both NG and CT infections will be low, but that much can be learned from the positive cases in terms of risk factors and optimal timing of screening. Further, the feasibility of screening in the third trimester will offer options for future guidelines.

ELIGIBILITY:
Inclusion criteria:

* all consecutive prenatal patients attending the obstetrical clinic at St. Michael's Hospital for a six-month period from May 1, 2016 to November 1, 2016, inclusive.

Exclusion criteria:

* none.

Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Pregnant women
Study Population: All consecutive prenatal patients attending the obstetrical clinic at St. Michael's Hospital for a six-month period from May 1, 2016 to November 1, 2016, inclusive.
Sampling Method: Probability Sample
Enrollment: 1691 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2019-02 (Actual); Study Completion 2019-02 (Actual)

PRIMARY OUTCOMES:
Rates of N. gonorrhoeae and C. trachomatis in the first trimester | first trimester (1-12 weeks gestation)
  To examine the incidence rates of N. gonorrhoeae and C. trachomatis in the first trimester of the obstetrical population at St. Michael's Hospital
Rates of N. gonorrhoeae and C. trachomatis in the third trimester | third trimester (29-40 weeks gestation)
  To examine the incidence rates of N. gonorrhoeae and C. trachomatis in the third trimester of the obstetrical population at St. Michael's Hospital

SECONDARY OUTCOMES:
Physician compliance with screening guidelines | first trimester (1-12 weeks gestation) and third trimester (29-40 weeks gestation)
  Assessment of physician compliance with Canadian screening and treatment guidelines which specify screening at first and third trimester

CONTACTS AND LOCATIONS:
Overall Officials: Mark Yudin, MD, Principal Investigator — Unity Health Toronto

IPD SHARING:
Plan to Share IPD: No